CLINICAL TRIAL: NCT05823090
Title: Light Therapy for Depression in Adolescent Outpatients: A Placebo lead-in Clinical Trial
Brief Title: Light Therapy for Depression in Adolescent Outpatients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Rachel Ballard, Physician, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-4706
Record Dates: First submitted 2023-03-27; First posted 2023-04-21 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Depression; Adolescent - Emotional Problem
Keywords: light therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: placebo lead-in open trial
Masking Description: Participants were blinded as to the type of light they received from the BLT device.
  Participants were assessed by both a blinded and non-blinded investigator. The blinded investigator assigned the Clinical Global Impressions Severity and Improvement Scales. The non-blinded investigator made clinical decisions regarding the BLT dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Bright light therapy (Experimental): Eligible participants were provided a light box and an actigraphy wrist-watch and given instructions on the use of each. The light therapy dosing protocol was planned as follows: Weeks 0-2, 50 lux dim red light (DRL) x 15 30 minutes/day; weeks 3-4, 10,000 lux x 15 minutes/day; weeks 5-6, 10,000 lux x 30 minutes/day; weeks 6-8, 10,000 lux x 45 minutes/day. At week 2, the study coordinator dispensed the 10,000 lux BLT unit (and picked up the DRL box) and the actigraphy watch. Participants and their parent/guardian met with 2 study clinicians at the end of each 2-week period. One study clinician, who was blinded to the participant's light box use, conducted a brief interview regarding mood, safety and functioning and side effects. The other study clinician subsequently met with the participant to review safety, side effects and response and made recommendations on duration and timing of light box use based on level of improvement and any barriers to use.
  Interventions: Device: light box (Carex DayLight Classic Model)

INTERVENTIONS:
Device: light box (Carex DayLight Classic Model) — The active light box is a white fluorescent 4000 Kelvin unit that emits 10,000 lux and measures 33cm x 40cm. The placebo box emits 50 lux dim red light and appears identical to the active unit. Subjects were instructed to position themselves 30-36 cm from the box with their faces fully exposed to the light. The actigraphy device is a Phillips Spectrum Plus Actigraphy watch which collects activity level and sleep information along with multiple light measurements and wearer adherence.

SUMMARY:
The goal of this placebo lead-in clinical trial was to test bright light therapy (BLT) in adolescents with depression. The main question[s] it aimed to answer were:

1. characterize and define facilitators/barriers to treatment with BLT in adolescents);
2. evaluate the acceptability and feasibility of outpatient BLT in a dose titration protocol;
3. establish an effective, safe and tolerable light dose.

DETAILED DESCRIPTION:
This outpatient study was performed at Ann & Robert H. Lurie Children's Hospital of Chicago. The Institutional Review Boards (IRB) of Lurie Children's Hospital and Northwestern University, Feinberg School of Medicine approved the protocol. Participants were recruited through partnering community pediatric practices (namely Lake Forest Pediatrics). Primary care pediatricians referred potential participants with depression and elevated scores on youth screening measures, Patient Health Questionnaire-9 (≥ 9) or PHQ-2 (≥ 3), without endorsed suicidality.

Light Therapy Protocol with Placebo Lead-in. Eligible participants were provided a light box and an actigraphy wrist watch and given instructions on the use of each. The active light box (Carex DayLight Classic Model) is a white fluorescent 4000 Kelvin unit that emits 10,000 lux and measures 33cm x 40cm. The placebo box emits 50 lux dim red light and appears identical to the active unit. Dim red light was selected because the illumination is a plausible placebo in clinical trials of BLT for depressive disorders and produces negligible effects on circadian rhythms and mood responses. Subjects were instructed to position themselves 30-36 cm from the box with their faces fully exposed to the light. The actigraphy device is a Philips Spectrum Plus actigraphy watch which collects activity level and sleep information along with multiple light measurements and wearer adherence. The light therapy dosing protocol was planned as follows: Weeks 0-2, 50 lux dim red light (DRL) x 30 minutes/day; weeks 3-4, 10,000 lux x 15 minutes/day; weeks 5-6, 10,000 lux x 30 minutes/day; weeks 6-8, 10,000 lux x 45 minutes/day. At week 2, the study coordinator (KJ) dispensed the 10,000 lux BLT unit (and picked up the dim red light box) and the actigraph watch. Participants and their parent/guardian met with 2 study clinicians at the end of each 2-week period. One study clinician (RB or JP), who was blinded to the participant's light box use, conducted a brief interview regarding mood, safety and functioning, and assigned a Clinical Global Impressions Scale-Severity (CGI-S). The other study clinician (DKS) subsequently met with the participant to review safety, side effects and response and made recommendations on duration and timing of light box use based on level of improvement and any barriers to use. Thus, some patients did not receive the above dosing schedule. After the 8-week active study period, participants who had symptom remission were given the option to keep the light box and continue use. A treatment summary and ongoing treatment recommendations were provided to all participant's primary care clinicians.

Adherence. The study coordinator made weekly calls/texts to participants to inquire about their daily exposure times and to encourage proper adherence. The constraints imposed upon adolescents by schools (early morning start times by 8:00 AM), bus commutes (pick up by 7:30 AM), after school activities and part-time jobs (landscaping etc.) are considerable. Knowing this and to avoid forcing adolescents to wake earlier than preferred (which can produce detrimental effects on adolescent sleep and mood) to use the study light box, participants agreed to initiate BLT exposure in the morning at awakening in accordance to the dosing protocol. At follow up visits, the non-blind clinician systematically explored whether morning use remained feasible and acceptable. If not, the clinician made informed clinical recommendations and recorded adjustments to the time-of-day of use (midday or afternoon) to ensure participants were able to consistently use the box. This strategy informed investigators and participants of the optimal timing of light exposure, increased adherence and strengthened the reliability of detecting response.

Actigraphic Assessments. Actigraphy using a wrist actigraph with a light sensor (Actiwatch Spectrum, Philips Respironics Healthcare, Bend, OR, USA) was used to measure a number of actigraphic-derived sleep, circadian, activity and light variables during the placebo and active light treatment phases.

ELIGIBILITY:
Inclusion Criteria:

* Participants with depression and elevated scores on youth screening measures, Patient Health Questionnaire-9 (PHQ-9 (≥ 9) or PHQ-2 (≥ 3).
* English-speaking primary caregiver legally able to provide consent and who could contribute weekly mood ratings.

Exclusion Criteria:

* Current or past diagnoses of bipolar disorder, moderate to severe autism, schizophrenia, or schizoaffective disorder, or intellectual disability; a major medical illness or ocular condition (e.g. glaucoma, retinal disease, macular degeneration) that would interfere with participation in the study; significant and imminent risk to self or to others; concurrent
* Recent (<4 months) medication or new (< 3 months) psychotherapy treatment for depression
* Current use of melatonin, beta-blockers, chloroquine, or regular non-steroidal anti-inflammatory agents, or St. John's Wort.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Adherence to BLT in adolescent outpatients with depression | 8 week study period
  Adherence to prescribed daily light box use measured by days used as a percentage of days prescribed.
Change in depression severity with dim red light (BLT placebo) | Baseline to study week 2
  Depression severity measured by child- and parent-report Short Mood and Feelings Questionnaire (score ranges from 0-26, with higher scores indicating worse outcome).
Change in depression severity with BLT | Study week 2 to study week 8
  Depression severity measured by child- and parent-report Short Mood and Feelings Questionnaire (score ranges from 0-26, with higher score indicating worse outcome).
Treatment emergent mania with dim red light (BLT placebo) in adolescent outpatients with depression | Baseline to study week 2
  Adverse event occurring during placebo phase as monitored by the parent-reported Child Mania Rating Scale (score range 0-30, with higher scores indicating worse outcomes).
Treatment emergent mania with BLT in adolescent outpatients with depression | Study week 2 to study week 8
  Adverse event occurring during BLT as monitored by the parent-reported Child Mania Rating Scale (score range 0-30, with higher scores indicating worse outcomes).
Treatment emergent suicidality with dim red light (BLT placebo) in adolescent outpatients with depression | Baseline to study week 2
  Adverse event occurring during placebo phase as monitored by the patient-reported Columbia Suicide Severity Rating Scale (3 questions; any "yes" answer indicates need for further clinical assessment).
Treatment emergent suicidality with BLT in adolescent outpatients with depression | Study week 2 to study week 8
  Adverse event occurring during BLT as monitored by the patient-reported Columbia Suicide Severity Rating Scale (3 questions; any "yes" answer indicates need for further clinical assessment).
Treatment emergent adverse events with dim red light (BLT placebo) in adolescent outpatients with depression | Baseline to study week 2
  Adverse event occurring during placebo phase as monitored by the and patient-reported Systematic Assessment for Treatment Emergent Effects (SAFTEE, modified, 26 items; range for any item 1-5 with 5 indicating worse outcome).
Treatment emergent adverse events with BLT in adolescent outpatients with depression | Study week 2 to study week 8
  Adverse event occurring during BLT as monitored by the and patient-reported Systematic Assessment for Treatment Emergent Effects (SAFTEE, modified, 26 items; range for any item 1-5 with 5 indicating worse outcome).

SECONDARY OUTCOMES:
Change in anxiety with BLT | Baseline to study week 8
  Anxiety severity measure by child- and parent-report Scale of Child Anxiety Related Disorders scale (score ranges from 0-82, with higher scores indicating worse outcomes).
Sleep efficiency and sleep onset latency with changing dose of BLT | Continuously through the 8-week study period
  sleep efficiency and sleep onset latency measured by actigraphy

CONTACTS AND LOCATIONS:
Locations (1):
- Rachel Ballard, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share individual participant data with other researchers.

REFERENCES:
- [Background] Oren DA, Brainard GC, Johnston SH, Joseph-Vanderpool JR, Sorek E, Rosenthal NE. Treatment of seasonal affective disorder with green light and red light. Am J Psychiatry. 1991 Apr;148(4):509-11. doi: 10.1176/ajp.148.4.509. PMID 2006698
- [Background] Sit DK, McGowan J, Wiltrout C, Diler RS, Dills JJ, Luther J, Yang A, Ciolino JD, Seltman H, Wisniewski SR, Terman M, Wisner KL. Adjunctive Bright Light Therapy for Bipolar Depression: A Randomized Double-Blind Placebo-Controlled Trial. Am J Psychiatry. 2018 Feb 1;175(2):131-139. doi: 10.1176/appi.ajp.2017.16101200. Epub 2017 Oct 3. PMID 28969438
- [Background] Wirz-Justice A, Bader A, Frisch U, Stieglitz RD, Alder J, Bitzer J, Hosli I, Jazbec S, Benedetti F, Terman M, Wisner KL, Riecher-Rossler A. A randomized, double-blind, placebo-controlled study of light therapy for antepartum depression. J Clin Psychiatry. 2011 Jul;72(7):986-93. doi: 10.4088/JCP.10m06188blu. Epub 2011 Apr 5. PMID 21535997
- [Background] Garbazza C, Cirignotta F, D'Agostino A, Cicolin A, Hackethal S, Wirz-Justice A, Cajochen C, Manconi M; "Life-ON" study group. Sustained remission from perinatal depression after bright light therapy: A pilot randomised, placebo-controlled trial. Acta Psychiatr Scand. 2022 Oct;146(4):350-356. doi: 10.1111/acps.13482. Epub 2022 Aug 3. PMID 35876837
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941